CLINICAL TRIAL: NCT05356780
Title: Predictability of Orthodontic Tooth Movement With Invisalign Aligners: Effect of Treatment Design and Operator Experience
Brief Title: Predictability of Orthodontic Tooth Movement With Invisalign Aligners
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Tommaso Castroflorio, Principal investigator, University of Turin, Italy
Other Study IDs: 157/2020
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Tooth Crowding; Malocclusion; Malocclusion, Angle Class II; Malocclusion, Class I/II
Keywords: Biomechanics; Aligner orthodontics; Adult patients; Orthodontic Tooth Movement predictability
MeSH Terms: conditions — Malocclusion; Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Expert operators
  Interventions: Device: Aligner
- Post-graduate students
  Interventions: Device: Aligner

INTERVENTIONS:
Device: Aligner — A method of straightening teeth without fixed braces

SUMMARY:
Together with the increased adult patient demand for orthodontic treatment and the push toward increasingly personalized treatment, technology developments have resulted in a growing worldwide demand for clear aligners, to the point that they are now an essential part of any orthodontic practice.

Despite the widespread use of the technique, the existing literature about reliability of orthodontic tooth movement with Invisalign aligners seems not encouraging. Several papers have demonstrated that what is virtually planned is not what is clinically achievable. However, it should be considered that clear aligner orthodontics techniques are customized not only for the patients but for orthodontists too. Therefore, virtual treatment plan design, in terms of attachments' design and placement, orthodontic tooth movement (OTM) staging and aligner deformation overengineering, or in other words aligners biomechanics knowledge, plays a crucial role in defining the quality of the orthodontic treatment with Invisalign aligners.

Based on these considerations the present study was designed to answer two research-clinical questions: 1) which are the less predictable orthodontic movements with Invisalign aligners when the treatment plan is designed by expert operators? and 2) which is the impact of the orthodontist experience, in terms of patient motivation, on the predictability of orthodontic tooth movement with Invisalign aligners? To answer those questions, the predictability of OTM in a sample of Invisalign patients treated by expert operators was compared with the predictability of OTM in a sample treated by post-graduate students.

The null hypothesis for question 1 is that all the prescribed orthodontic tooth movements are predictable, while the null hypothesis for question 2 is that the reliability of orthodontic tooth movement is not affected by operator experience.

98 patients (31 M, 67 F; mean age 28 ± 12 years) were selected among those in treatment at the Department of Orthodontics of the University of Turin, which is the coordinating center, and at 5 private orthodontics offices across Italy. The inclusion criteria for practitioners were as follows: orthodontist with huge and renewed experience in Invisalign treatments; has the ability to scan plaster model or to collect intraoral scans and upload (via internet) the files obtained to a central repository; affirms that the practice can devote sufficient time in patient scheduling to allow focused recording of all data required for the study; and does not anticipate retiring, selling the practice, or moving during the study. Signed, written informed consent was required before inclusion in the trial.

All participants included in this prospective observational study had Class I or mild Class II malocclusion with mild to moderate crowding or spacing in the maxillary and mandibular dental arches (nonextraction cases). Interproximal enamel reduction was performed as prescribed in each patient's virtual treatment plan.

The average treatment time was 10 ± 5 months. The sample considered a total of 2716 teeth that were analyzed overlapping the real post-treatment .stl file obtained with the final intra-oral scan to the planned post-treatment .stl file obtained exporting the final stage of the virtual setup.

Every virtual treatment plan was designed by orthodontists with a huge and renewed experience in Invisalign treatments. While in the private practices the treatment was directly conducted by 5 expert orthodontist (mean age 45.6 ± 8.2) who controlled the patient at every appointment, in the University setting the treatment was conducted by 5 post-graduate students at the last year of their program (mean age 26.4± 1.4). Control appointments were fixed at 6 weeks interval in both the University and the private settings.

Posttreatment digital models and final virtual treatment plan models were exported from ClinCheck® software as stereolithography files and subsequently imported into Geomagic Qualify software (3D Systems(r), Rock Hill, South Carolina, USA), in order to compare individual tooth positions between digital models of each patient. The dental arches were superimposed using the landmark-based method and the surface-based method (Best Fit Alignment). So that the differences between the tooth positions could be calculated, 3 reference planes were identified on the virtual treatment plan model. Differences between the actual treatment outcome and the predicted outcome were calculated and tested for statistical significance for each tooth in the mesial-distal, vestibular-lingual, and occlusal-gingival directions, as well as for angulation, inclination, and rotation. Differences greater than 0.5 mm for linear measurements and 2° for angular measurements were considered clinically significant. In addition, the statistical significance of categorical variables was tested for each previously calculated difference in tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* complete permanent dentition, with the exception of third molars;
* Invisalign treatment in both arches;
* active tooth movements programmed at the standard rate recommended by the Align Tech technician;
* no intermediate corrections or additional aligners;
* aligners change every 7 to 14 days;
* good patient compliance.

Exclusion Criteria:

* need for oral surgery or dental restorations;
* failure to complete the initial series of aligners;
* combo treatments (i.e. combination of aligners with any other orthodontic appliance);
* poor patient cooperation;
* previous orthodontic treatment;
* presence of prosthetic restorations and/or periodontal problems
* signs and/or symptoms of temporomandibular disorders.

Ages: 11 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: orthodontic patients affering to the department of Turin and patients affering to 5 private orthodontics offices across Italy
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Predictable orthodontic movements with Invisalign aligners | 1 month
  Differences between the actual treatment outcome and the predicted outcome were calculated and tested for statistical significance for each tooth in the mesial-distal, vestibular-lingual, and occlusal-gingival directions, as well as for angulation, inclination, and rotation. Differences greater than 0.5 mm for linear measurements and 2° for angular measurements were considered clinically significant. In addition, the statistical significance of categorical variables was tested for each previously calculated difference in tooth movement.

SECONDARY OUTCOMES:
The impact of the orthodontist experience, on the predictability of orthodontic tooth movement with Invisalign aligners | 1 months
  The predictability of OTM in a sample of Invisalign patients treated by expert operators was compared with the predictability of OTM in a sample treated by post-graduate students

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Castroflorio, DDS, PhD, Study Chair — Department of Orthodontics of the University of Turin
Locations (1):
- Department of Orthodontics of the University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: No